CLINICAL TRIAL: NCT06026072
Title: Prospective Validation of the CLAD Score in Patients Admitted to an Emergency Facility for Renal Colic Pain
Brief Title: Validation of the CLAD Score Ifor Renal Colic Pain
Acronym: CLAD-V
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC31/21/0124; 2021-A00807-34 (Other: ID-RCB)
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Renal Colic
MeSH Terms: conditions — Renal Colic

STUDY DESIGN:
Intervention Model Description: The doctor in charge of the patient will have to examine him and take care of him according to the service protocol. He will also completed the CLAD-V score and gives his intuition on the surgical outcome of the patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CLAD-V (Other): All patient with renal colic will be eligible. The CLAD-V score will fills by the doctor and seven days after the patient will call back to know if he had a surgical intervention or no.
  Interventions: Other: CLAD-V SCORE

INTERVENTIONS:
Other: CLAD-V SCORE — the CLAD-V score is measured by the doctor during the emergency take care. After 7 days the patient will be call back to compare the prediction of CLAD-V score and the reality of surgical intervention or no.

SUMMARY:
Renal colic is a frequent reason for recourse representing 1 to 2% of emergency room admissions.

This study would validate the performance of the CLAD score in predicting the need for surgical management within 7 days of patients admitted to the emergency department for renal colic pain.

DETAILED DESCRIPTION:
Renal colic is a frequent reason for recourse representing 1 to 2% of emergency room admissions. It results clinically in a lumbo-abdominal pain syndrome radiating into the genitals. The origin of this pain is the tensioning of the urinary tract, most frequently by a lithiasis creating a transient obstruction

Toulouse medical team has developed the "Complicated uroLithiasis and Alternative Diagnosis" (CLAD) score, which predicts the risk of requiring surgery within 7 days of admission of patients to the emergency room for renal colic

The aim of this study is to validate this CLAD-V score by collecting the elements of the CLAD score and the clinician's intuition is made available to practitioners in the emergency department.

All patients presenting to the emergency room for renal colic pain are eligible. The doctor in charge of the patient will have to examine him and take care of him according to the service protocol. The doctor must then complete the questionnaire provided.

A reminder of the patient on D7 is carried out to collect information on the need for surgery after the emergency or not.

Each center ensures inclusions and reminders on D7 and will only transmit the database

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to the emergency room for suspected renal colic
* Patient not objecting to participation

Exclusion Criteria:

* Patients unable to express their non-objection
* Pregnant women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
CLAD-V performance | 7 days
  Validate the performance of the CLAD score in predicting the need for surgical management within 7 days of patients admitted to the emergency department for renal colic pain

CONTACTS AND LOCATIONS:
Overall Officials: Frederic BALEN, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, Haute-Garonne, France